CLINICAL TRIAL: NCT02437214
Title: Randomized Single Blinded Clinical Trial on Effects of Nursery Songs in Infants and Young Children's Anxiety Prior and During Head CT
Brief Title: Music to Decrease Pain and Anxiety During Head CTs Performed at the PEds ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Weiss (Other)
Responsible Party: Sponsor-Investigator, Steven Weiss, Professor of Emergency Medicine, University of New Mexico
Organization: University of New Mexico (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07-030
Record Dates: First submitted 2015-04-16; First posted 2015-05-07 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Anxiety Disorder of Childhood or Adolescence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of music for anxiety in children (Experimental): Children in the Exp group received the usual medical care in combination with the intervention. The intervention was started by the patients nurse without the knowledge of the research associate. In the intervention group, music was played until the CT scan was completed.
  Interventions: Other: Use of music for anxiety in children
- Control (No Intervention): Children in the Con group received the usual medical care without listening to the music intervention.

INTERVENTIONS:
Other: Use of music for anxiety in children — The "Baby Go to Sleep" CD played a combination of the sound of an actual human heartbeat and children's songs. The concept behind the "Baby Go to Sleep" CD is to blend heart beat sounds, which are known to be calming to infants and children, with children's music. The basic principles of relaxation were incorporated in the arrangements of heartbeat and children's songs, ie: simplicity, repetition, predictability, and simple symmetry (short repeated patterns). The adult human heart in the "Baby Go to Sleep" CD was recorded from the chest and set in consistent tempos for each song ranging from 62 to 78 beats per minute(BPM). The sound of the heartbeat continued between and during songs. Tempo changes occurred between each song.
  Arms: Use of music for anxiety in children

SUMMARY:
A single blinded controlled trial to determine if an intervention of listening to nursery songs with integrated heart beat sounds results in changes in anxiety level in infants and young children less than four years of age in an emergent setting.

DETAILED DESCRIPTION:
This study is a prospective cohort with a randomized single-blinded intervention with convenience sampling design. Our pediatric emergency medicine department (PED) treats nearly 2,500 patients between 1 and 3 years of age annually in 2008-10 and is a regional referral center for specialty care for our state. All data is collected in the PED between May 2008 and July 2010.

One PED examination room is designated as the study room. The music was stored on an ipod played in a portable speaker. The music is from the Compact Disk(CD), "Baby Go to Sleep." This is a commercially available CD.23 The "Baby Go to Sleep" Compact Disk played a combination of the sound of an actual human heartbeat and children's songs. Tempo changes occurred between each song. During the study, the initial three nursery rhymes were played.

The principal investigator's research associates recruit all patients up to 3 years of age presenting to the PED during the hours they were available. Once situated in the room, children both in the control and experimental group received the usual medical care including the evaluation by attending physician to determine if head CT would be performed or not. After subjects were determined to need a head CT by the attending physicians, they were randomly assigned to either the Control(Con) or experimental(Exp) group. Children in the Con group received the usual medical care while children in the Exp group received the usual medical care in combination with the intervention. The intervention was started by the patients nurse without the knowledge of the research associate. In the intervention group, music was played until the CT scan was completed. Research associates rated children's anxiety levels using a visual analogue scale(VAS) and Modified Ramsay Sedation Scale(MRSS) before children were transferred to radiology department for head CT then after children was laid down to go through head CT. Researchers associates were blinded to group by wearing headphones that were tested to ensure that they could not hear whether or not music was playing during the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* We sampled all children up to ages 3 years who present to the PED during the hours that the research assistant was present to collect data.

Exclusion Criteria:

* All children requiring trauma room care were excluded because they were not able to move to the study's examination room after triage (their care will be completed in the trauma room). Children with hearing deficit and those who are unable to move to the designated examination room for other reasons including needing oxygen and cardiopulmonary monitoring were excluded as well. The patients were also excluded if we were unable to track their results or chart at final review of patient data.

Ages: 1 Month to 36 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale of anxiety | up to 10 minutes
  A 100 mm scale completed by the research associate relating the degree of infant anxiety

SECONDARY OUTCOMES:
Modified Ramsey Sedation Scale | up to 10 minutes
  A validated 1-6 likert scale for measuring degree of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weiss, MD, Study Director — University of New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park G, Weiss SJ, Repar P. Randomized single-blinded clinical trial on effects of nursery songs for infants and young children's anxiety before and during head CT. Am J Emerg Med. 2016 Mar;34(3):663. doi: 10.1016/j.ajem.2015.12.049. Epub 2015 Dec 21. No abstract available. PMID 26782796
- [Derived] Park G, Weiss SJ, Repar P. Randomized single-blinded clinical trial on effects of nursery songs for infants and young children's anxiety before and during head computed tomography. Am J Emerg Med. 2015 Oct;33(10):1477-82. doi: 10.1016/j.ajem.2015.07.045. Epub 2015 Jul 29. PMID 26314215